CLINICAL TRIAL: NCT00247546
Title: Prevention of Falls and Injurious Falls Among Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital District of Satakunta (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 02032002
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-09

CONDITIONS: Falls; Accidental Falls
Keywords: Falls; Accidental falls; Prevention; Aged; Multifactorial trial

INTERVENTIONS:
Behavioral: Multifactorial prevention

SUMMARY:
The aim of this study is to describe and analyse the effects of multifactorial trial on the incidence of falls and injurious falls and on different risk factors of falling among the home-dwelling aged.

DETAILED DESCRIPTION:
The aims of the study:

1. To implement a program for the prevention of falls and injurious falls.
2. To describe the structure and activities of the fall prevention program implemented among the aged who are living in their own home, have at least moderate cognitive abilities, have fallen during previous 12 months and are 65 years of age or older. A further aim is to describe the frequency of participation according to age, gender, residence, health and physical condition.
3. To describe the effects of prevention on primary risk factors of falling such as muscle strength, balance, eye sight, medications, depression and home hazards in relation to age, gender, health and physical condition.
4. To describe and assess the effects of prevention on the incidence of falls and injurious falls.
5. To assess the effects of prevention on physical, cognitive and psychosocial functional abilities, quality of life and use of health and social services and deaths.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* home-dweller
* having fallen at least once during the previous 12 months
* at least moderate cognitive abilities (MMSE over 17)
* able to walk 10 metres independently

Exclusion Criteria:

* MMSE under 17

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 592
Dates: Start 2003-03; Study Completion 2005-03

PRIMARY OUTCOMES:
Incidence of falls and injurious falls

SECONDARY OUTCOMES:
Risk factors of falling
Functional abilities
Quality of life
Use of health and social services
Deaths

CONTACTS AND LOCATIONS:
Overall Officials: Sirkka-Liisa Kivelä, Professor, Study Director — The Hospital District of Satakunta
Locations (1):
- The Hospital District of Satakunta, Pori, Finland

REFERENCES:
- [Derived] Salminen M, Vahlberg T, Kivela SL. The long-term effect of a multifactorial fall prevention programme on the incidence of falls requiring medical treatment. Public Health. 2009 Dec;123(12):809-13. doi: 10.1016/j.puhe.2009.10.018. PMID 19958918